CLINICAL TRIAL: NCT05600244
Title: Comparison of Pericapsular Nerve Group Block, Quadratus Lumborum Block and Lumbar Erector Spinae Plane Block for Acute Pain Management in Total Hip Surgery: A Randomized Clinical Trial
Brief Title: PENG vs. QLB vs. Lumbar ESPB in Total Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKSU 50-9-21
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Total Hip Surgery; Pericapsular Nerve; Quadratus Lumborum; ESPB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG block Technique (Experimental): Patients will receive ultrasound-guided Pericapsular Nerve Group Block using 30 ml bupivacaine 0.25%.
  Interventions: Procedure: PENG block Technique
- Lumbar ESPB Technique (Experimental): Patients will receive lumbar erector spinae plane block using 30 ml bupivacaine 0.25%
  Interventions: Procedure: Lumbar ESPB Technique
- Transmuscular QLB-t block Technique (Experimental): Patients will receive transmuscular quadratus lumborum block using 30 ml bupivacaine 0.25%
  Interventions: Procedure: Transmuscular QLB-t block Technique

INTERVENTIONS:
Procedure: PENG block Technique — A linear probe will be used. Puncture will be performed in a lateromedial direction until the needle tip reached the plane between the iliopsoas tendon and periosteum and between the anterior inferior iliac spine and iliopubic eminence. After a negative aspiration test, 30 ml of bupivacaine 0.25% will be injected in the plane beneath the iliopsoas muscle
  Arms: PENG block Technique
Procedure: Lumbar ESPB Technique — Using the out-plane technique, a 22G/80-mm block needle will be advanced until it reached the transverse process. 0.5-1 ml of the prepared local anesthetic solution, 30 ml bupivacaine 0.25% will be administered leading to hydrodissection to confirm the correct location. The needle will be repositioned by pulling back a few millimeters if resistance occurs when administering local anesthetic . All local anesthetic will be administered to this location between the transverse process and the erector spinae muscle
  Arms: Lumbar ESPB Technique
Procedure: Transmuscular QLB-t block Technique — A convex transducer will be placed in the transverse plane on the flank of the patient cranial to the iliac crest. The 4th lumbar vertebral transverse process, erector spinae muscles, psoas muscle, transverse abdominis muscle, internal and externa oblique muscles, and the quadratus lumborum muscle will be identified. A 15 cm 22G insulated needle will be inserted on the posterior corner of the transducer. 30 ml bupivacaine 0.25% will be administered between the quadratus lumborum and psoas muscles into the fascial plane.
  Arms: Transmuscular QLB-t block Technique

SUMMARY:
The aim of this study is to compare between Pericapsular Nerve Group Block, Erector Spinae Plane Block and Quadratus Lumborum Block for managing acute postoperative pain in patients undergoing total hip surgeries under spinal anesthesia.

DETAILED DESCRIPTION:
Total hip surgeries are one of the most common major orthopedic procedures to improve patient's functional status and quality of life. However, despite these advantages, the immediate postoperative period can be associated with severe pain that delays mobilization and increases hospital stay and the risk of thromboembolic events.

Various methods are used for postoperative pain management. Intravenous opioid agents are among them, but they may cause undesirable side effects, such as respiratory depression, sedation, constipation, allergic reaction, nausea, and vomiting. Thus, alternative techniques are preferred.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Both genders
* Body mass index < 40 kg/m^2
* American Society of Anesthesiologists (ASA) physical status I-III
* Posted for total hip surgeries under spinal anesthesia

Exclusion Criteria:

* The presence of contraindications or allergy to local anesthetic agents
* Chronic use of opioids or corticosteroids
* Infection at the puncture site
* Coagulopathy
* Psychiatric disorders (dementia or cognitive impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Total amount of rescue analgesia | 24 hours postoperatively
  Total amount of rescue analgesia in the form of morphine will be recorded

SECONDARY OUTCOMES:
First analgesic request | 24 hours Postoperatively
  The time to first request of rescue analgesia will be recorded
Pain level | 48 hours Postoperatively
  Pain level will be evaluated using numeric rating analogue scale (NRS), which ranges from 0 to 10 points, with 0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Adverse events | 48 hours Postoperatively
  Adverse events will be recorded (e.g., nausea, vomiting, hypotension and bradycardia)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Fouad Algyar, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available under a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study